CLINICAL TRIAL: NCT05392712
Title: Ultra-sensitive Magnetocardiography in the Accurate Identification of Severe Coronary Lesions and Myocardial Necrosis
Brief Title: Magnetocardiography in the Accurate Identification of Severe Coronary Lesions and Myocardial Necrosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Weifang People's Hospital (Other); Linyi People's Hospital (Other); Jining First People's Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Chongqing Emergency Medical Center (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); First People's Hospital of Hangzhou (Other); Qianfoshan Hospital (Other); Weihai Central Hospital (Other); Heze Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: QLEmer-Magneto 1
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-05

CONDITIONS: Chest Pain, Acute Coronary Syndrome, Myocardial Infarction
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- healthy volunteers (Other)
  Interventions: Device: Magnetometer
- Chest pain patients who will undergo CAG or CTA (Experimental)
  Interventions: Device: Magnetometer
- AMI patients (Experimental)
  Interventions: Device: Magnetometer

INTERVENTIONS:
Device: Magnetometer — inspection equipment for magnetocardiography

SUMMARY:
Magnetocardiography (MCG) is a promising noninvasive and accurate method for detecting myocardial ischemia. Although progress has been made in this area, there is a lack of studies using up-to-date examination instruments for the calibration of MCG analysis. This is a prospective single-center study aiming to build accurate analytical models of MCG to detect coronary lesions and myocardial necrosis. Coronary lesions are measured by coronary angiography (CAG) or coronary CTA, and are defined by both the stenosis degree and the computer-simulated fraction flow reserve. Myocardial necrosis is examined and quantified by cardiac MR. Healthy volunteers, chest pain patients who will receive CAG or CTA examination, and patients with acute myocardial infarction will be enrolled in this study.

ELIGIBILITY:
For healthy volunteers:

Inclusion Criteria:

1. Age 18-79 years old;
2. No history of cardiovascular disease (coronary heart disease, structural heart disease, arrhythmia, heart failure, stroke, pulmonary embolism, aortic dissection, etc.), no cardiovascular risk factors (hypertension, diabetes, hyperlipidemia). For people over 65 years old, those with hypertension or hyperlipidemia, but with well-controlled blood pressure and lipid levels, taking no more than 2 drugs, and echocardiography showing no left ventricular hypertrophy, can be included;
3. The electrocardiogram is normal, and the cardiac ultrasound is basically normal in the past 1 year (mild valvular regurgitation can be included).
4. Sign the informed consent.

Exclusion Criteria:

1. Those who with acute or chronic respiratory diseases;
2. Those who with obvious abnormality of liver or kidney function;
3. Those who with endocrine diseases such as abnormal thyroid function;
4. Those who with anemia or other blood diseases;
5. Those who with connective tissue diseases (lupus erythematosus, rheumatoid arthritis, dermatomyositis, polyarteritis nodosa, etc.);
6. Those who are obese (BMI>30kg/cm2) or underweight (BMI<18kg/cm2);
7. Those who with malignant tumors;
8. Those who with infectious diseases or infectious diseases;
9. Those who with trauma or physical disability;
10. Those who with psychological or mental illness such as depression;
11. Those who are professional athletes, pregnant or breastfeeding women, alcoholics;
12. Those who are unable to perform magnetocardiography examination due to claustrophobia, etc., or those who fail to receive magnetocardiography examination;
13. Due to various reasons such as allergy to contrast agents, metal implants in vivo that are prohibited from performing 1.5T MRI (such as prostheses or steel plates implanted in orthopaedics, uterine contraceptive device) and other reasons, those who cannot or fail to cooperate with the corresponding research requirements.

For chest pain patients who will undergo CAG or CTA:

Inclusion Criteria:

1. Age 18-79 years old;
2. Those with chest pain symptoms, diagnosed or highly suspected by the attending doctor or above as stable angina pectoris (SA), unstable angina pectoris (UA), non-ST segment elevation myocardial infarction (NSTEMI), ST segment elevation myocardial infarction (STEMI), and plan to receive CAG or coronary CTA;
3. Sign the informed consent.

Exclusion Criteria:

1. Patients with known structural heart disease such as cardiomyopathy and valvular disease;
2. Patients with arrhythmias such as atrial fibrillation, supraventricular tachycardia, and atrioventricular block that have not returned to normal;
3. History of other cardiovascular diseases such as pulmonary embolism and aortic dissection;
4. Patients with connective tissue diseases (lupus erythematosus, rheumatoid arthritis, dermatomyositis, polyarteritis nodosa, etc.) combined with cardiac complications;
5. Obvious abnormal thyroid function, severe anemia or other blood diseases and other diseases that obviously affect the circulating blood supply;
6. Obese (BMI>30kg/cm2) or underweight (BMI<18kg/cm2);
7. Patients with malignant tumors;
8. Professional athletes, pregnant or breastfeeding women, alcoholics;
9. Acute diseases or critical illnesses in other systems, such as acute or severe respiratory diseases, abnormal liver function or renal function, etc.;
10. Patients with infectious diseases or infectious diseases;
11. Those who are unable or fail to perform magnetocardiography due to claustrophobia, physical impairment, etc.;
12. Unable to or fail to cooperate with the corresponding research requirements.

For AMI patients:

Inclusion Criteria:

1. Age 18-79 years old;
2. The attending doctor or above has diagnosed the patient as acute myocardial infarction (NSTEMI, STEMI), the condition of whom is relatively stable, and CMR examination is feasible after evaluation.
3. Sign the informed consent.

Exclusion Criteria:

1. Patients with known structural heart disease such as cardiomyopathy and valvular disease;
2. Patients with arrhythmias such as atrial fibrillation, supraventricular tachycardia, and atrioventricular block that have not returned to normal;
3. History of other cardiovascular diseases such as pulmonary embolism and aortic dissection;
4. Patients with connective tissue diseases (lupus erythematosus, rheumatoid arthritis, dermatomyositis, polyarteritis nodosa, etc.) combined with cardiac complications;
5. Obvious abnormal thyroid function, severe anemia or other blood diseases and other diseases that obviously affect the circulating blood supply;
6. Obese (BMI>30kg/cm2) or underweight (BMI<18kg/cm2);
7. Patients with malignant tumors;
8. Professional athletes, pregnant or breastfeeding women, alcoholics;
9. Acute diseases or critical illnesses in other systems, such as acute or severe respiratory diseases, abnormal liver function or renal function, etc.;
10. Patients with infectious diseases or infectious diseases;
11. Those who are unable or fail to perform magnetocardiography due to claustrophobia, physical impairment, etc.;
12. Due to various reasons such as allergy to contrast agents, metal implants in vivo that are prohibited from performing 1.5T MRI (such as prostheses or steel plates implanted in orthopaedics, uterine contraceptive device) and other reasons, those who cannot or fail to cooperate with the corresponding research requirements.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of MCG to detect coronary lesion | 24 hours
  To establish an algorithm model of MCG in detecting coronary lesion and to assess the sensitivity and specificity of the above model in detecting coronary lesion. Coronary lesion is measured by degree of stenosis via CAG/CTA and computer-simulated fraction flow reserve via QFR/CTFFR.
Accuracy of MCG to detect myocardial necrosis | 24 hours
  To establish an algorithm model of MCG in detecting myocardial necrosis and to assess the sensitivity and specificity of this model in detecting myocardial necrosis, which is measured via cardiac MR.

SECONDARY OUTCOMES:
Accuracy of MCG to detect the localization of coronary lesion | 24 hours
  To build up an algorithm model of MCG in detecting the localization of coronary lesion. Assess the sensitivity and specificity of this model to detect the main vessels where the lesion locates.
Accuracy of MCG to detect the zone of myocardial necrosis | 24 hours
  To establish an algorithm model of MCG to detect the infarct zone of the heart. Assess the sensitivity and specificity of this model to detect the location of myocardial necrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Yuguo Chen, Dr, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China